CLINICAL TRIAL: NCT04174664
Title: Comparison of Different Functional Capacity Tests in Cystic Fibrosis Patients With Acute Pulmonary Exacerbation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Kübra Kılıç, MSc, PT, Hacettepe University
Other Study IDs: GO 19/817
Record Dates: First submitted 2019-11-13; First posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Cystic Fibrosis in Children; Exercise Capacity
Keywords: pulmonary exacerbation
MeSH Terms: interventions — Exercise Test; Respiratory Function Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 1-minute sit to stand test — Childrens will complete 1-minute sit to stand test and 3 minute step test and quality of life questionnaire.
  Other Names: 3-minute step test; Quality of life; pulmonary function test

SUMMARY:
The aim of this study to investigate and compare functional capacity with different tests and to evaluate the relationship between functional capacity and quality of life during acute pulmonary exacerbation in children with cystic fibrosis.

Exercise tests associated with prognostic values in CF patients and decreased exercise capacity has been correlated with a reduction in health-related quality of life. Pulmonary functions, functional capacity and quality of life will examine in this study.

DETAILED DESCRIPTION:
This study will be participated children with cystic fibrosis who will diagnosed acute pulmonary exacerbation. Patients' pulmonary function test, functional capacity will be assess and record at hospital admission and hospital discharge and outpatient clinic control. Quality of life will be evaluated at only outpatient clinic control .

Pulmonary function test will be assessed with spirometry, functional capacity will be evaluated with 1-minute sit to stand test and 3-minute step test. And quality of life will be evaluated Cystic Fibrosis Questionnaire-Revised (CFQ-R).

ELIGIBILITY:
Inclusion Criteria:

* Childrens with CF diagnosed between 7-18 years of age and hospitalized due to acute pulmonary exacerbation will be included in the study.The diagnosis of acute pulmonary exacerbation will be established by Fuchs criteria.

Exclusion Criteria:

* Patients with allergic bronchopulmonary aspergillosis (ABPA) who were treated with systemic steroid therapy and noninvasive mechanical ventilation support will not be included in the study.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Acute pulmonary exacerbation in childrens with cystic fibrosis diagnosed according to Fuchs criteria.
Sampling Method: Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
1 minute sit to stand test (STS) repetitions | November 2019- January 2021
  number of STS completed at hospital admissions, hospital discharge and outpatient time
3 minute step test | November 2019- January 2021
  number of completed step at hospital admissions, hospital discharge and outpatient time
pulmonary functions | November 2019- January 2021
  pulmonary functions assessment via spirometry
Quality of life assesment | November 2019- January 2021
  Cystic Fibrosis Questionnaire-Revised (CFQ-R) included 4 different age. These versions are teen/adult version,child version,parent version for children, preschool version. Scores range from 0 to 100, with higher scores indicating better health. This questionnaire will be filled only once.

SECONDARY OUTCOMES:
Maximal heart rate | November 2019- January 2021
  maximal heart rate during 3-minute step test
Heart rate | November 2019- January 2021
  difference pre and post test heart beat number
oxygen saturation | November 2019- January 2021
  difference pre and post test percentage of oxygen saturation
dyspnea | November 2019- January 2021
  difference pre and post test breathlessness with Visual Analogue Scale (VAS).Scores range from 0 to 10, with higher scores indicating worse outcome.
quadriceps fatigue | November 2019- January 2021
  difference pre and post test quadriceps fatigue with Visual Analogue Scale (VAS).Scores range from 0 to 10, with higher scores indicating worse outcome.
fatigue | November 2019- January 2021
  difference pre and post test fatigue with Visual Analogue Scale (VAS).Scores range from 0 to 10, with higher scores indicating worse outcome.
hospitalization frequency | 1 year
  number of hospitalization per year

CONTACTS AND LOCATIONS:
Overall Officials: Naciye Vardar-Yagli, PhD, Study Director — Hacettepe University; Deniz Inal-Ince, Professor, Study Chair — Hacettepe University; Melda Saglam, PhD, Study Chair — Hacettepe University; Ebru Yalcin, Professor, Study Chair — Hacettepe University; Dilber Ademhan-Tural, MD, Study Chair — Hacettepe University; Kubra Kilic, MSc, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided